CLINICAL TRIAL: NCT03897439
Title: Individualizing Pharmacotherapy: A Novel Optimization Strategy to Increase Smoking Cessation in the African American Community
Brief Title: Individualizing Pharmacotherapy for African American Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nikki Nollen, PhD, MA, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study0000142310; R01DA046576 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Varenicline; Bupropion

STUDY DESIGN:
Intervention Model Description: African American smokers randomized to OPT (n=196) will receive high intensity smoking cessation counseling, nicotine patch (NP), and up to two pharmacotherapy optimizations [varenicline (VAR), bupropion (BUP) plus NP] based on verified smoking status at Weeks 2 and 6.
  African American smokers randomized to enhanced UC (n=196) will receive the same high intensity counseling and NP with no optimizations in pharmacotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (UC) (Active Comparator): 196 African American smokers will receive 12 weeks of smoking cessation counseling and 18 weeks of nicotine patch.
  Interventions: Drug: Nicotine patch
- Optimized Care (OPT) (Experimental): 196 African American smokers will receive 12 weeks of smoking cessation counseling. They will receive the nicotine patch and up to two pharmacotherapy adaptations (VAR, BUP+NP) based on verified smoking status at Weeks 2 and 6 for a total of 18 weeks of pharmacotherapy.
  Interventions: Drug: Nicotine patch; Drug: Varenicline Tartrate; Drug: Bupropion

INTERVENTIONS:
Drug: Nicotine patch — Participants will receive the 24-hour 21mg nicotine patch for up to 18 weeks of treatment.
  Other Names: Nicoderm
Drug: Varenicline Tartrate — VAR will be dispensed 0.5 mg once daily on Days 1-3, 0.5 mg twice daily on Days 4-7, and 1 mg twice daily from Day 8 through the end of treatment.
  Other Names: Chantix
  Arms: Optimized Care (OPT)
Drug: Bupropion — BUP will be dispensed 150 mg once daily on Days 0-3 and then 150 mg twice daily from Day 4 through optimization or the end of treatment.
  Other Names: Zyban; Wellbutrin
  Arms: Optimized Care (OPT)

SUMMARY:
Improving cessation outcomes for African American smokers through the use of novel, empirically-based strategies is a national health priority. In the vast majority of smoking cessation studies and in clinical practice, when smokers are provided a medication to help them quit, they are expected to continue that medication regardless of how well it is working. This study will assess whether African Americans smokers respond better if they continue with a single treatment or if their treatment is changed when that treatment is not working.

DETAILED DESCRIPTION:
The objective of this study is to examine the efficacy of optimized (OPT) versus enhanced usual care (UC) treatment for smoking cessation. African American smokers randomized to OPT (n=196) will receive high intensity smoking cessation counseling, nicotine patch (NP), and up to two pharmacotherapy optimizations [varenicline (VAR), bupropion (BUP) plus NP, ] based on verified smoking status at Weeks 2 and 6. African American smokers randomized to enhanced UC (n=196) will receive the same high intensity counseling and NP with no optimizations in pharmacotherapy. Pharmacotherapy and counseling in both groups will last for 18 weeks with long-term follow-up through Week 26. The primary outcome is biochemically-verified smoking status at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic African American
* ≥ 18 years of age
* Smoke 5-30 cigarettes per day (CPD)
* Daily cigarette smoker
* Smoked at current rate for > 6 months
* Verified smoker (CO > 5 ppm)
* Functioning telephone
* Interested in quitting smoking
* Willing to take NP, VAR , and/or BUP+NP for 18 weeks and complete all study visits

Exclusion Criteria:

* Use of non-cigarette tobacco products in past 30 days
* Medical contraindications to NP, BUP, or VAR: unstable cardiac condition (e.g., unstable angina or AMI) cardiac event, or stroke in the past 4 weeks; renal impairment; medications contraindicated ; history of clinically significant allergic reactions; history of epilepsy, seizure, head trauma, psychosis, bipolar disorder, eating disorder; unstable panic disorder or depression; active suicidal ideation; treatment for alcohol or drug dependence in the past year
* Use of pharmacotherapy in the month prior to enrollment
* Pregnant, contemplating getting pregnant, or breastfeeding
* Unstable housing (e.g., street, shelter)
* Plans to move from Kansas City during the treatment and follow-up phase
* Another household member enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nollen, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Swope Health Central, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambart LM, Cox LS, Mayo MS, Brown AR, Leavens ELS, Ahluwalia JS, Nollen NL. Change in Cigarette, Other Tobacco Product, and Cannabis Use Among Individuals Who Used or Did Not Use Cannabis During a Smoking Cessation Trial. Nicotine Tob Res. 2025 Aug 22;27(9):1641-1646. doi: 10.1093/ntr/ntaf045. PMID 39976595
- [Derived] Nollen NL, Ahluwalia JS, Mayo MS, Ellerbeck EF, Leavens ELS, Salzman G, Shanks D, Woodward J, Greiner KA, Cox LS. Multiple Pharmacotherapy Adaptations for Smoking Cessation Based on Treatment Response in Black Adults Who Smoke: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317895. doi: 10.1001/jamanetworkopen.2023.17895. PMID 37338906
- [Derived] Nollen NL, Cox LS, Mayo MS, Ellerbeck EF, Arnold MJ, Salzman G, Shanks D, Woodward J, Greiner KA, Ahluwalia JS. Protocol from a randomized clinical trial of multiple pharmacotherapy adaptations based on treatment response in African Americans who smoke. Contemp Clin Trials Commun. 2022 Nov 5;30:101032. doi: 10.1016/j.conctc.2022.101032. eCollection 2022 Dec. PMID 36387983

RESULTS

PARTICIPANT FLOW:
Period: Randomization (Week 0)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 196 | 196
Started on Nicotine Patch | 196 | 196
Completed | 196 | 196
Not Completed | 0 | 0
Period: Optimization Point 1 (Week 2)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 187 (9 participants were lost to follow-up between period 1 and 2) | 187 (9 participants were lost to follow-up between period 1 and period 2)
Stayed on Nicotine Patch | 187 | 61
Adapted to VAR | 0 | 126
Completed | 187 | 187
Not Completed | 0 | 0
Period: Optimization Point 2 (Week 6)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 178 (9 participants were lost to follow-up between period 2 and period 3.) | 173 (14 participants were lost to follow-up between period 2 and period 3.)
Stayed on Nicotine Patch | 178 | 52
Stayed on VAR | 0 | 25
Adapted to Varenicline | 0 | 9
Adapted to BUP + Nicotine Patch | 0 | 87
Completed | 178 | 173
Not Completed | 0 | 0
Period: Primary Endpoint (Week 12)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 174 (4 participants were lost to follow-up between period 3 and period 4.) | 165 (8 participants were lost to follow-up between period 3 and period 4.)
Completed | 174 | 165
Not Completed | 0 | 0
Period: End of Treatment (Week 18)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 170 (4 participants were lost to follow-up between period 4 and period 5.) | 163 (2 participants were lost to follow-up between period 4 and period 5.)
Completed | 170 | 163
Not Completed | 0 | 0
Period: End of Study (Week 26)
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Started | 162 (8 participants were lost to follow-up between period 5 and period 6.) | 162 (1 participant was lost to follow-up between period 5 and period 6.)
Completed | 162 | 162
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: 196 African American smokers will receive 12 weeks of smoking cessation counseling and 18 weeks of nicotine patch.
  Nicotine patch: Participants will receive the 24-hour 21mg nicotine patch for up to 18 weeks of treatment.
- Optimized Care: 196 African American smokers will receive 12 weeks of smoking cessation counseling. They will receive the nicotine patch and up to two pharmacotherapy adaptations (VAR, BUP+NP) based on verified smoking status at Weeks 2 and 6 for a total of 18 weeks of pharmacotherapy.
  Nicotine patch: Participants will receive the 24-hour 21mg nicotine patch for up to 18 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Optimized Care | Total
Number analyzed (Participants) | 196 | 196 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (11.5) | 52.3 (11.7) | 52.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 114 | 224
  Male | 86 | 82 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 196 | 196 | 392
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 196 | 196 | 392
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 196 | 196 | 392
Cohabitation Status; Married/Living with partner [Count of Participants; unit: Participants] | 62 | 54 | 116
Employment Status; Not currently employed [Count of Participants; unit: Participants] | 107 | 124 | 231
Education Level; some college or technical school [Count of Participants; unit: Participants] | 86 | 101 | 187
Has Health Insurance [Count of Participants; unit: Participants] — Do you have health insurance that pays for most of your medical care (yes, no)?
  Participants | 138 | 124 | 262
% with a Federal Poverty Level <=100% [Count of Participants; unit: Participants] — Federal poverty level is determined by a combination of total income and number of people in the household. Thresholds are defined annually by HHS.
  Participants | 87 | 99 | 186
Housing; Own a home [Count of Participants; unit: Participants] | 36 | 29 | 65
Cigarettes per day in the past 7 days [Mean (Standard Deviation); unit: cigarettes per day] | 13.3 (7.3) | 12.2 (6.9) | 12.8 (7.1)
Menthol smoker [Count of Participants; unit: Participants] | 172 | 173 | 345

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically Verified Smoking Abstinence at Week 12
Description: Biochemically verified 7-day point prevalence abstinence defined as smoking zero cigarettes at Week 12 visit. This will evaluate the short-term efficacy of optimized pharmacotherapy for smoking cessation in African American smokers.
Time Frame: Week 12
Population: Intent to treat with missing treated as smokers
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Number analyzed (Participants) | 196 | 196
Participants | 23 | 34

2. Secondary Outcome: Number of Participants With Biochemically Verified Smoking Abstinence at Week 18
Description: Biochemically verified 7-day point prevalence abstinence defined as smoking zero cigarettes at Week 18 visit. This will evaluate the end-of-treatment efficacy of optimized pharmacotherapy for smoking cessation in African American smokers
Time Frame: Week 18
Population: Intent to treat with missing treated as smokers
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Number analyzed (Participants) | 196 | 196
Participants | 31 | 32

3. Secondary Outcome: Number of Participants With Biochemically Verified Smoking Abstinence at Week 26
Description: Biochemically verified 7-day point prevalence abstinence defined as smoking zero cigarettes at Week 26 visit. This will evaluate the long-term efficacy of optimized pharmacotherapy for smoking cessation in African American smokers
Time Frame: Week 26
Population: Intent to treat with missing treated as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
Number analyzed (Participants) | 196 | 196
Participants | 26 | 24

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through Week 18.
Description: Adverse event data was collected at each follow-up timepoint with a series of global side effect questions and a prompt to report an adverse events. Events are reported by group, overall (OPT, UC) , and not per intervention within group (e.g., optimized care: NP, optimized care: VAR, optimized care: BUP + NP) because many participants in OPT received all interventions and it is not possible to separate the adverse events they experienced during each of the interventions they received.
Arm/Group | Usual Care (UC) | Optimized Care (OPT)
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/196
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/196
Other Adverse Events (participants affected / at risk) | 25/196 | 19/196
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (UC) (N=196) | Optimized Care (OPT) (N=196)
Redness/swelling/rash on the skin (General disorders) | 25 | 19
Sleeping Problems (General disorders) | 3 | 14
Nausea or Vomiting (Gastrointestinal disorders) | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03897439/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT03897439/ICF_001.pdf